CLINICAL TRIAL: NCT00357682
Title: A Phase III, Randomized, Study of Aspirin and Esomeprazole Chemoprevention in Barrett's Metaplasia
Acronym: AspECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000491649; OCTO-003 (Other: Oncology Clinical Trials Office); 2004-003836-77 (EudraCT Number); ISRCTN85156844 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2018-08

CONDITIONS: Esophageal Cancer; Precancerous Condition
Keywords: esophageal cancer; Barrett's esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Precancerous Conditions; Barrett Esophagus | interventions — Esomeprazole; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): 20mg Esomeprazole
  Interventions: Drug: Esomeprazole
- Arm B (Experimental): 80mg Esomeprazole
  Interventions: Drug: Esomeprazole
- Arm C (Experimental): 20mg Esomeprazole + 300mg Aspirin
  Interventions: Drug: Esomeprazole; Drug: Aspirin
- Arm D (Experimental): 80mg Esomeprazole + 300mg Aspirin
  Interventions: Drug: Esomeprazole; Drug: Aspirin

INTERVENTIONS:
Drug: Esomeprazole — 20mg per day
  Other Names: Nexium
  Arms: Arm A; Arm C
Drug: Esomeprazole — 80mg per day
  Other Names: Nexium
  Arms: Arm B; Arm D
Drug: Aspirin — 300mg per day
  Arms: Arm C; Arm D

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of esomeprazole and aspirin may prevent esophageal cancer in patients with Barrett's metaplasia. It is not yet known whether esomeprazole is more effective with or without aspirin in preventing esophageal cancer in patients with Barrett's metaplasia.

PURPOSE: This randomized phase III trial is studying esomeprazole with or without aspirin to compare how well they work in preventing esophageal cancer in patients with Barrett's metaplasia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

* To assess whether intervention with aspirin results in a decreased rate of all causes of mortality or conversion rate from Barrett's metaplasia to adenocarcinoma or high grade dysplasia.
* To assess whether high dose PPI (protein pump inhibitor) therapy results in a decreased rate of all causes of mortality or conversion rate from Barrett's metaplasia to adenocarcinoma or high grade dysplasia.

SECONDARY OBJECTIVES

* To assess whether intervention with aspirin results in decreased high-grade dysplasia, in decreased all cause mortality, in decreased oesophageal cancer incidence and in decreased cause-specific mortality when each is considered separately
* To assess whether intervention with high dose PPI results in decreased high-grade dysplasia, in decreased all cause mortality, in decreased oesophageal cancer incidence and in decreased cause-specific mortality when each is considered separately
* To assess whether there are clinical and molecular risk factors which can be identified in BM (Barrett's Metaplasia) for the development of BA.
* To assess the cost effectiveness of aspirin and/or PPI treatment in the prevention of BA.
* To assess whether intervention with PPI and/or aspirin induces changes in the expression of molecular markers for BA.
* To investigate new genes important in the progression of BA, as a unique tissue bank will be available with a complete endoscopic, histological, physiology and pharmaceutical history.
* To assess inherited genetic factors for predisposition to oesophagitis above BM, BM, LGD HGD and BA.
* To assess what the biological risk factors are for cardiac disease and aspirin resistance.
* To assess gender differences in outcomes.

Cancer Research UK approved the study in 2003 for a 10 year period to run from 1st January 2005 to 31st December 2014. Funding is renewable annually and is dependent on a satisfactory review by an independent committee.

An application for a funding extension was made to CRUK 18 months before the end of the grant and the funding was extended to 31Aug2018.

A total of 2557 patients have been accrued for this study in the UK.

ELIGIBILITY:
INCLUSION CRITERIA

1. Aged ≥18 years.
2. Circumferential Barrett's metaplasia of at least 1cm in length (≥C1M1) or a tongue of Barrett's metaplasia of at least 2cm in length (≥C0M2) (irrespective of the presence now or historically of histologically proven intestinal metaplasia).
3. Able to give written informed consent.
4. WHO performance status of 0 or 1 i.e. fully active and self-caring.

EXCLUSION CRITERIA

1. High grade dysplasia or carcinoma at enrolment.
2. Medical conditions which would make completing endoscopies or completing the trial difficult including:

   1. Frequent transient ischaemic attacks (3 or more) or severe cerebral vascular accident in the previous 6 months*
   2. Severe respiratory disease with arterial oxygen saturation less 90% at rest
   3. Severe ischaemic heart disease (exercise tolerance less than 100 yards or life expectancy < 4 years) or myocardial infarction in the previous 3 months
   4. Severe inflammatory bowel disease requiring at least one hospital admission of 5 days in the last year or bowels open > 6 times/day * Patients answering yes to criterion a. were eligible for the PPI-only (non-aspirin) arms of the trial
3. Continuous/frequent non-steroidal anti-inflammatory drug use or COX-2 inhibitors (more than 60 days per year in total).
4. Patients with absolute contraindications to PPIs, aspirin or their excipients i.e. allergies, ulcers, renal impairment or use of oral anticoagulants.
5. Pregnant or lactating women will not undergo endoscopy and may be given dispensation to stop drug therapy for a year. This should be discussed with the Trial Office.

If a patient was suitable for inclusion but later becomes unsuitable this should be discussed with the Trial Office before they are withdrawn. Only in exceptional circumstances should patients not be followed up i.e. withdrawal of consent or current life threatening disease with poor outcome and therefore unable to tolerate endoscopy. In these circumstances patients should be followed up in outpatient clinics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2557 (Actual)
Dates: Start 2005-03-10 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Jankowski, MD, Principal Investigator — National Institute for Health and Care Excellence

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jankowski JAZ, de Caestecker J, Love SB, Reilly G, Watson P, Sanders S, Ang Y, Morris D, Bhandari P, Brooks C, Attwood S, Harrison R, Barr H, Moayyedi P; AspECT Trial Team. Esomeprazole and aspirin in Barrett's oesophagus (AspECT): a randomised factorial trial. Lancet. 2018 Aug 4;392(10145):400-408. doi: 10.1016/S0140-6736(18)31388-6. Epub 2018 Jul 26. PMID 30057104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2557 eligible participants were recruited across from 4th March 2005 to 25th February 2009. There were 84 centres across England, Scotland, Wales, and Northern Ireland, and one in McMaster Health Sciences Centre, Hamilton, ON, Canada.
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C | Arm D
Started | 705 | 704 | 571 | 577
Completed | 364 | 394 | 320 | 312
Not Completed | 341 | 310 | 251 | 265
Not completed — Did not receive allocated Treatment | 10 | 9 | 9 | 10
Not completed — Withdrew consent | 6 | 6 | 5 | 5
Not completed — Lost to Follow-up | 39 | 33 | 26 | 35
Not completed — Adverse Event | 24 | 32 | 22 | 27
Not completed — Physician Decision | 32 | 20 | 24 | 30
Not completed — Patient decision | 73 | 80 | 51 | 59
Not completed — Other reason | 157 | 130 | 114 | 99

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Arm D | Total
Number analyzed (Participants) | 699 | 698 | 566 | 572 | 2535
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 495 | 494 | 429 | 418 | 1836
  >=65 years | 204 | 204 | 137 | 154 | 699
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 136 | 118 | 124 | 513
  Male | 564 | 562 | 448 | 448 | 2022
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: First Event of Death, Oesophageal Adenocarcinoma, High Grade Dysplasia
Description: Death is recorded on a continuous basis through reporting from trial sites. Oesophageal adenocarcinoma is recorded through endoscopies taken every two years or ad-hoc at clinician decision High Grade Dysplasia is recorded through endoscopies taken every two years or ad-hoc at clinician decision
Time Frame: Events are assessed from the date of randomisation to the end of study which can be patient withdrawal, loss to follow up or study end (8 years or 10 years from randomisation, depending on consent)
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Groups:
- Aspirin: Subjects randomised to receive 300mg daily aspirin
- No Aspirin: Subjects randomised to receive no aspirin
- Low Dose PPI: Subjects randomised to receive 20mg daily PPI
- High Dose PPI: Subjects randomised to receive 80mg daily PPI
Arm/Group | Aspirin | No Aspirin | Low Dose PPI | High Dose PPI
Number analyzed (Participants) | 1138 | 1142 | 1265 | 1270
Participants | 127 | 154 | 174 | 139
Statistical Analysis 1: Comparison: Low Dose PPI vs High Dose PPI; Accelerated Failure Time (AFT) analysis comparing time to primary event in low dose PPI (20mg) patients to high dose PPI (80mg) patients. Included in AFT model are stratification factors (Barrett's length, age group and presence of baseline intestinal metaplasia) and aspirin randomisation group; Test type: Superiority — 5% significance level is considered statistically significant; p = 0.068, Accelerated Failure Time; Time Ratio = 1.24, 95% CI 2-sided [0.98 to 1.57]
Statistical Analysis 2: Comparison: Aspirin vs No Aspirin; Accelerated Failure Time (AFT) analysis comparing time to primary event in aspirin patients to non-aspirin patients. Included in AFT model are stratification factors (Barrett's length, age group and presence of baseline intestinal metaplasia) and PPI randomisation group; Test type: Superiority — 5% significance level is considered statistically significant; p = 0.037, Accelerated Failure Time; Time Ratio = 1.27, 95% CI 2-sided [1.01 to 1.58]

2. Secondary Outcome: All Cause Mortality
Description: Accelerated Failure Time (AFT) analysis comparing time to all cause mortality in low dose PPI (20mg) patients to high dose PPI (80mg) patients and in aspirin patients to non-aspirin patients. Included in AFT model are stratification factors (Barrett's length, age group and presence of baseline intestinal metaplasia) and aspirin randomisation group.
Time Frame: Through study completion, an average of 8.9 years.
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | No Aspirin | Low Dose PPI | High Dose PPI
Number analyzed (Participants) | 1138 | 1142 | 1265 | 1270
Participants | 73 | 90 | 105 | 79
Statistical Analysis 1: Comparison: Low Dose PPI vs High Dose PPI; All recordings of death, regardless of the cause are used in this analysis and both PPI groups are compared; Test type: Superiority — 5% significance level is considered statistically significant; p = 0.039, Accelerated Failure Time; Time Ratio = 1.36, 95% CI 2-sided [1.01 to 1.82]
Statistical Analysis 2: Comparison: Aspirin vs No Aspirin; There are 163 deaths in the aspirin comparison with all-cause mortality as the endpoint. Median follow-up is 8.9 years IQR: (8.2 , 10.0) Range: (0 , 11.5); Test type: Superiority — 5% significance level is considered statistically significant; p = 0.159, Accelerated Failure Time; Time Ratio = 1.25, 95% CI 2-sided [0.92 to 1.70]

3. Secondary Outcome: Adenocarcinoma Oesophageal Cancer
Description: Number of aspirin and non-aspirin patients and low dose PPI and high dose PPI patients with adenocarcinoma oesophageal cancer
Time Frame: Assessed every 2 years through study completion, an average of 8.9 years
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | No Aspirin | Low Dose PPI | High Dose PPI
Number analyzed (Participants) | 1138 | 1142 | 1265 | 1270
Participants | 35 | 35 | 41 | 40
Statistical Analysis 1: Comparison: Low Dose PPI vs High Dose PPI; There are 81 diagnoses in the PPI dose comparison with adenocarcinoma oesophageal cancer as the endpoint. Median follow-up is 8.7 years IQR: (8.1 , 9.9); Test type: Superiority — 5% significance level is considered statistically significant; p = 0.864, Accelerated Failure Time; Time Ratio = 1.04, 95% CI 2-sided [0.67 to 1.61]
Statistical Analysis 2: Comparison: Aspirin vs No Aspirin; There are 70 diagnoses of adenocarcinoma in the aspirin comparison. Median follow-up is 8.8 years, IQR: (8.1 , 10), Range: (0 , 11.5); Test type: Superiority — 5% significance level is considered statistically significant; p = 0.921, Accelerated Failure Time; Time Ratio = 1.02, 95% CI 2-sided [0.64 to 1.64]

4. Secondary Outcome: High Grade Dysplasia
Description: Diagnosis of high grade dysplasia is compared in aspirin and non-aspirin trial patients, and in high dose PPI and low dose PPI patients.
Time Frame: High Grade Dysplasia is assessed every two years through study completion, an average of 8.9 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin | No Aspirin | Low Dose PPI | High Dose PPI
Number analyzed (Participants) | 1138 | 1142 | 1265 | 1270
Participants | 37 | 55 | 59 | 44
Statistical Analysis 1: Comparison: Low Dose PPI vs High Dose PPI; There are 103 such diagnoses in the PPI dose comparison. Median follow-up is 8.7 years IQR: (8.1 , 9.9) Range: (0 , 11.48); Test type: Superiority — 5% significance level is considered statistically significant; p = 0.119, Accelerated Failure Time; Time Ratio = 1.36, 95% CI 2-sided [0.92 to 2.02]
Statistical Analysis 2: Comparison: Aspirin vs No Aspirin; There are a total of 92 conversions to HGD in the aspirin comparison. Median follow-up is 8.8 years IQR (8.1 , 10.0) Range (0 , 11.5); Test type: Superiority — 5% significance level is considered statistically significant; p = 0.053, Accelerated Failure Time; Time Ratio = 1.51, 95% CI 2-sided [1.00 to 2.29]

ADVERSE EVENTS:
Time Frame: Adverse event monitoring started from the time the patient commenced study medication until 30 days after stopping trial medication (an average of 8.9 years).
Arm/Group | Aspirin | No Aspirin | Low Dose PPI | High Dose PPI
All-Cause Mortality (participants affected / at risk) | 73/1138 | 90/1142 | 105/1265 | 79/1270
Serious Adverse Events (participants affected / at risk) | 340/1138 | 378/1142 | 359/1265 | 359/1270
Other Adverse Events (participants affected / at risk) | 0/1138 | 0/1142 | 0/1265 | 0/1270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin (N=1138) | No Aspirin (N=1142) | Low Dose PPI (N=1265) | High Dose PPI (N=1270)
Hematoma (Vascular disorders) | 0 | 2 | 0 | 2
Hypertension (Vascular disorders) | 1 | 1 | 2 | 0
Hypotension (Vascular disorders) | 3 | 0 | 1 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 2 | 1 | 1
Ruptured aortic arch aneurism (Vascular disorders) | 2 | 1 | 1 | 2
Thromboembolic event (Vascular disorders) | 10 | 12 | 11 | 11
Vasculitis (Vascular disorders) | 1 | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 1 | 4
Brain cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 10 | 8 | 8
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Gastric - Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Laryngeal - Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 12 | 12 | 10
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 3 | 2
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1 | 2
Metastatic cancer unknown origin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 2
Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 2
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3 | 0
Oesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 5 | 1
Oral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 2 | 3
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 3 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 11 | 6 | 13
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 5 | 2
Skin cancer melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 3
Skin cancer non-melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 3 | 1
Testicular cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 1 | 0 | 2
Anaphylaxis (Immune system disorders) | 0 | 1 | 0 | 1
Autoimmune disorder (Immune system disorders) | 0 | 2 | 1 | 1
Fetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0
Fever (General disorders) | 1 | 1 | 0 | 2
Flu like symptoms (General disorders) | 0 | 1 | 0 | 1
Injection site reaction (General disorders) | 0 | 1 | 1 | 0
Localized edema (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 19 | 19 | 14 | 24
Pain (General disorders) | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 4 | 2 | 0 | 6
Mania (Psychiatric disorders) | 0 | 1 | 1 | 0
Psychosis (Psychiatric disorders) | 1 | 1 | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 2 | 0 | 3
Accidental death (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Alcohol abuse (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 4 | 4 | 5 | 3
Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Cholecystectomy procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 4 | 5 | 6
Fracture (Injury, poisoning and procedural complications) | 11 | 9 | 9 | 11
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 10 | 8 | 5
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 3 | 2 | 3 | 2
Ruptured spleen (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 4 | 3 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0
GGT increased (Investigations) | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0
Vitamin B12 deficiency (Investigations) | 0 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 7 | 6 | 3 | 10
Aortic dissection (Cardiac disorders) | 0 | 1 | 0 | 1
Aortic stenosis (Cardiac disorders) | 1 | 1 | 1 | 1
Aortic valve disease (Cardiac disorders) | 1 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 8 | 10 | 11 | 7
Atrial flutter (Cardiac disorders) | 1 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 1 | 2 | 1
Cardiac arrest (Cardiac disorders) | 2 | 3 | 4 | 1
Cardiomyopathy (Cardiac disorders) | 2 | 4 | 2 | 4
Chest pain (Cardiac disorders) | 8 | 15 | 10 | 13
Heart failure (Cardiac disorders) | 5 | 5 | 6 | 4
Myocardial infarction (Cardiac disorders) | 24 | 24 | 23 | 25
Pericardial effusion (Cardiac disorders) | 1 | 1 | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 1 | 1 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 6 | 1 | 4 | 3
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 2 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 2 | 11 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 4
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 6 | 9 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 6 | 5 | 8 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 6 | 5 | 5
Intracranial hemorrhage (Nervous system disorders) | 5 | 5 | 5 | 5
Ischemia cerebrovascular (Nervous system disorders) | 18 | 17 | 18 | 17
Memory impairment (Nervous system disorders) | 1 | 1 | 2 | 0
Motor neurone disease (Nervous system disorders) | 0 | 1 | 0 | 1
Multiple system atrophy (Nervous system disorders) | 0 | 1 | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 2 | 3 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 1 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0
Spasticity (Nervous system disorders) | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 3 | 4 | 5 | 2
Transient ischemic attacks (Nervous system disorders) | 10 | 8 | 7 | 11
Vasovagal reaction (Nervous system disorders) | 0 | 1 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 1 | 0 | 2
Vitreous hemorrhage (Eye disorders) | 2 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 1 | 3
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 6 | 10 | 6
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Bloating (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Cameron Ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 0 | 0 | 3
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 2 | 3 | 2 | 3
Constipation (Gastrointestinal disorders) | 2 | 3 | 2 | 3
Diverticulitis (Gastrointestinal disorders) | 4 | 5 | 5 | 4
Duodenal hemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 2 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 3 | 1 | 3 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 3 | 2 | 4 | 1
Oesophageal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 4 | 2 | 3 | 3
Gastritis (Gastrointestinal disorders) | 2 | 2 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 7 | 2 | 6
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 | 0 | 2 | 1
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Ileal obstruction (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ischaemic Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Mallory-Weiss tear (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 9 | 8 | 9 | 8
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 3 | 3 | 4
Vomiting (Gastrointestinal disorders) | 6 | 1 | 2 | 5
Acute kidney injury (Renal and urinary disorders) | 3 | 3 | 2 | 4
Chronic kidney disease (Renal and urinary disorders) | 1 | 3 | 2 | 2
Haematuria (Renal and urinary disorders) | 2 | 4 | 3 | 3
Renal calculi (Renal and urinary disorders) | 2 | 3 | 4 | 1
Renal colic (Renal and urinary disorders) | 1 | 4 | 4 | 1
Urinary retention (Renal and urinary disorders) | 3 | 5 | 3 | 5
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 1 | 1
Alcoholic Hepatitis (Hepatobiliary disorders) | 2 | 0 | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 13 | 9 | 12 | 10
Gallbladder necrosis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 2 | 2 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 4 | 3 | 4 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2
Cervical Spondylosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Hernia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 2
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Mortons neuroma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Tendon rupture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Goitre (Endocrine disorders) | 1 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 4 | 2 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 1
Anorectal infection (Infections and infestations) | 2 | 0 | 0 | 2
Appendicitis (Infections and infestations) | 3 | 2 | 0 | 5
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Bladder infection (Infections and infestations) | 0 | 2 | 2 | 0
Bone infection (Infections and infestations) | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 1 | 1 | 1
Enterocolitis infectious (Infections and infestations) | 9 | 9 | 8 | 10
Eye infection (Infections and infestations) | 1 | 0 | 1 | 0
Hepatic infection (Infections and infestations) | 1 | 0 | 0 | 1
Inner Ear Infection (Infections and infestations) | 0 | 1 | 0 | 1
Intestinal parasite (Infections and infestations) | 1 | 0 | 1 | 0
Joint infection (Infections and infestations) | 0 | 2 | 1 | 1
Kidney infection (Infections and infestations) | 0 | 2 | 1 | 1
Lung infection (Infections and infestations) | 25 | 31 | 28 | 28
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Prostate infection (Infections and infestations) | 0 | 1 | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 1 | 0 | 1
Salivary gland infection (Infections and infestations) | 1 | 0 | 1 | 0
Scrotal infection (Infections and infestations) | 2 | 1 | 0 | 3
Sepsis (Infections and infestations) | 1 | 2 | 2 | 1
Skin infection (Infections and infestations) | 7 | 14 | 9 | 12
Soft tissue infection (Infections and infestations) | 1 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 2 | 0 | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 11 | 4 | 8 | 7
Wound infection (Infections and infestations) | 1 | 6 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-01-26): https://cdn.clinicaltrials.gov/large-docs/82/NCT00357682/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT00357682/SAP_001.pdf